CLINICAL TRIAL: NCT00757393
Title: Growth Hormone Therapy and Bone Quality in Pediatric Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Etienne Sochett, Staff Endocrinologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000012269
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Osteoporosis
Keywords: Growth hormone; Pediatrics; Vitamin D; Calcium; Exercise
MeSH Terms: conditions — Osteoporosis; Motor Activity | interventions — Vitamin D; Calcium; Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D + Calcium + Exercise program
- 2 (Experimental)
  Interventions: Drug: Vitamin D + Calcium + Exercise program + Humatrope

INTERVENTIONS:
Dietary Supplement: Vitamin D + Calcium + Exercise program — Subjects is this arm of the study will receive a) a supplementation with vitamin D3, 1000 IU daily b) a dietary calcium intake set at DRI for age and a supplement used as needed to meet the requirement and c) a weight bearing exercise program appropriate for the underlying medical condition
  Arms: 1
Drug: Vitamin D + Calcium + Exercise program + Humatrope — Subjects in this arm will receive the same as those in arm 1 as well as Humatrope by subcutaneous infection 7 days a week at a dose of 0.05 mg.kg/day.
  Other Names: Growth Hormone
  Arms: 2

SUMMARY:
The primary objective of this study is to test the hypothesis that growth hormone, administered daily by subcutaneous injection for 2 years will result in a significantly greater BMD Z-score over optimal standard therapy.

DETAILED DESCRIPTION:
Osteoporosis is a skeletal disorder characterized by a parallel loss of bone mineral and matrix which results in enhanced bone fragility and an increased risk of fractures. The associated fractures, and the morbidity and mortality that ensue, make osteoporosis a public health problem of enormous proportions. Clinical and research observations strongly suggest that most adult osteoporosis has its roots in childhood and have identified both genetic and environmental factors as central to the pathogenesis of this disorder.

Osteoporosis is not only a major public health problem in the adult population but is increasingly diagnosed during childhood. Most cases are secondary to chronic illnesses (secondary osteoporosis). In chronically ill children several factors, in addition to the underlying chronic illness itself, may predispose to either reduced bone mass or impairment of bone quality. Osteoporosis in the otherwise healthy child (primary osteoporosis) is generally classified as either osteogenesis imperfecta (OI) or juvenile idiopathic osteoporosis (JIO).

Optimizing Vitamin D and calcium intake as well as a weight bearing exercise program are central approaches in the prevention and treatment of osteoporosis. Despite increased awareness of this disorder in the pediatric population and more active implementation of these principles, an ever increasing number of children with osteoporosis present with symptomatic disease; that is progress to the stage of frequent peripheral fractures, vertebral compression fracture and/or deliberating pain. Bisphosphonates are often then added to the therapeutic regiment. However, it is widely acknowledged that little is currently known about the key factors that might predict the safe and effective use of these agents in this population.

Children whose bone biopsy results indicate an adynamic form of osteoporosis and who have low bone turnover markers make up a significant number of the children with symptomatic osteoporosis. Many of these patients have in addition growth failure (due to prolonged glucocorticoid usage and chronic illness) and some may have low growth hormone secretion. In this circumstance, the agent of choice would be an anabolic agent known to increase osteoblast activity, normalize histomorphometric parameters and improve bone quality. Unfortunately, one of the most promising of these agents, recombinant PTH (Teripeptide) is precluded from use in pediatric patients because of concerns regarding induction of osteosarcoma. It is unclear to what extent antiresorptive therapy might achieve these goals, although it has become the therapy of choice by default.

The Growth hormone (GH)/IGFI- axis plays a central role in longitudinal bone growth as well as in the acquisition and maintenance of bone mass in children. Studies, in both growth hormone excess and deficiency, suggest that growth hormone may be useful as an anabolic agent in children with osteoporosis. In acromegaly, bone turnover markers indicate activation of both osteoblasts and osteoclasts. Both markers correlate with circulating GH and IGF-1 levels. IGF-1 levels are increased in cortical bone suggesting that the anabolic actions of GH are mediated by local production. The impact on bone density in unclear, as some studies show no differences from healthy controls. However, other studies indicate an increase in cortical bone mass while trabecular mass appears to be unchanged or somewhat reduced. Furthermore rates appear not to be increased.

The Growth hormone (GH)/IGFI-axis plays a central role in the longitudinal bone growth as well as in the acquisition and maintenance of bone mass in children. Studies, in both growth hormone excess and deficiency, suggest that growth hormone may be useful as an anabolic agent in children with osteoporosis. Growth hormone deficiency (GHD) is recognized to result in reduced bone mass, decreased bone turnover markers, secondary osteoporosis and increased fracture rate. Epidemiological studies suggest that GHD alone may explain the increased fracture rate seen in these patients. Treatment of GHD patients with GH results in an increase in turnover markers. While short-term studies showed little improvement in bone mass, longer term studies with treatment periods of 2 years or more have shown significant increases in bone mass.

ELIGIBILITY:
Inclusion Criteria:

* Adynamic form of osteoporosis based on bone biopsy findings
* Age range 5-16 years
* Willingness to comply with the protocol
* Underlying primary disorder (when present) in a maintenance phase of treatment and the patient considered to be clinically stable

Exclusion Criteria:

* Previous treatment with an antiresorptive agent within 1 year of commencement of the study
* Unstable primary disorder (when present)
* Significant psychosocial difficulties that will likely preclude compliance with the protocol
* Any contraindication to the use of growth hormone
* Patients with severe osteoporosis and past medical history of malignancy

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2008-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Test the hypothesis that growth hormone administered daily by subcutaneous injection for 2 years will result in a significantly greater BMD Z-score over optimal standard therapy | 2 years

SECONDARY OUTCOMES:
Test the hypothesis that subcutaneous growth hormone administration will significantly improve and/or normalize baseline values of fracture frequency | 2 years
Test the hypothesis that subcutaneous growth hormone administration will significantly improve and/or normalize baseline values of bone histomorphometric measures osteoid volume, surface, and width | 2 years
Test the hypothesis that subcutaneous growth hormone administration will significantly improve and/or normalize baseline measures of bone quality | 2 years
Test the hypothesis that subcutaneous growth hormone administration will significantly improve and/or normalize baseline values of BMC corrected for height | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Sochett, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada